CLINICAL TRIAL: NCT06130826
Title: A Phase I Study of M5A-IL2 Immunocytokine Combined With Stereotactic Body Radiation Therapy (SBRT) in Patients With Metastatic Colorectal Cancer or CEA-Positive Metastatic Breast Cancer
Brief Title: Immune Response Activation for the Treatment of Unresectable Metastatic Colorectal Cancer or CEA Positive Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20510; NCI-2023-07592 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20510 (Other: City of Hope Medical Center); P30CA033572 (NIH); R01CA283603 (NIH)
Record Dates: First submitted 2023-10-20; First posted 2023-11-14 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Breast Carcinoma; Colorectal Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms | interventions — Biopsy; Specimen Handling; Immunotherapy; Adjuvants, Immunologic; Magnetic Resonance Spectroscopy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (SBRT, M5A-IL2 ICK) (Experimental): Patients undergo SOC SBRT over 3 fractions on days 1, 3, and 5, followed by M5A-ICK SC on days 8, 9, and 10 once daily for a single cycle on study. Patients undergo CT or PET/CT as well as blood sample collection throughout the trial. Patients may undergo magnetic resonance imaging or bone scan as clinically indicated on the trial. Additionally, patients may optionally undergo tissue biopsy during screening and on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Immunotherapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Immunotherapy — Receive M5A-IL2 ICK SC
  Other Names: Immunological; Immunological Therapy; Immunologically Directed Therapy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase I trial studies the side effects and best dose of M5A-IL2 immunocytokine (M5A-ICK) combined with stereotactic body radiation therapy (SBRT) and to see how well they work in treating patients with colorectal cancer or xarcinoembryonic antigen (CEA) positive breast cancer that cannot be removed by surgery (unresectable) or has spread from where it first started (primary site) to other places in the body (metastatic). Carcinoembryonic Antigen (CEA) is a protein that is present in most colorectal cancers and in many other cancers, such as breast cancer, as well. SBRT uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Cytokines are signaling proteins that help control inflammation in the body. They allow the immune system to mount a defense if germs or cancer or other substances that can make people sick enter the body. Interleukin-2 (IL-2) is a powerful cytokine able to regulate the immune responses that are important for anticancer immunity. Immunocytokines (also called antibody-cytokine fusion proteins) are small proteins that regulate the activity of immune cells. The M5A-IL2 immunocytokine (M5A-ICK) combines the cancer targeting features of the M5A antibody with the immune system regulation properties of the cytokine IL-2. Giving M5A-ICK in combination with standard of care (SOC) SBRT may work better in treating patients with unresectable metastatic colorectal cancer or CEA positive metastatic breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Identify the maximum tolerated dose (MTD) and recommend phase 2 dose (RP2D) and characterize toxicities associated with administration of the M5A-IL2 after fractionated SBRT.

SECONDARY OBJECTIVES:

I. Describe the therapeutic response to treatment of irradiated and unirradiated tumors per Criteria in Solid Tumors version 1.1 (RECIST v 1.1) guidelines.

II. Describe AEs by M5A-IL2 dose level, per Common Terminology Criteria for Adverse Events [CTCAE] version 5.0.

III. Describe the pharmacokinetics of M5A-IL2. IV. Describe the frequency of auto-antibody formation, overall and by dose of M5A-IL2.

EXPLORATORY OBJECTIVE:

I. If medically feasible, tumors targeted for SBRT will be biopsied pre-SBRT and 1-2 weeks post 3rd dose of M5A-IL2.

OUTLINE: This is a dose-escalation study of M5A-ICK.

Patients undergo SOC SBRT over 3 fractions on days 1, 3, and 5, followed by M5A-ICK subcutaneously (SC) on days 8, 9, and 10 once daily for a single cycle on study. Patients undergo computed tomography (CT) or positron emission tomography (PET)/CT as well as blood sample collection throughout the trial. Patients may undergo magnetic resonance imaging or bone scan as clinically indicated on the trial. Additionally, patients may optionally undergo tissue biopsy during screening and on study.

After completion of study treatment, patients are followed-up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have a diagnosis of metastatic colon or rectal or breast cancer that is pathology proven
* Patients should have a CEA producing colorectal cancer or breast cancer defined as a baseline CEA or prior documented CEA level exceeding 5 ng/ml or evidence of CEA staining by Immunohistochemistry (IHC)
* Patients should 18 years of age or older
* Patients are willing and capable to consent to study and to adhere with all elements of the study
* Patients who have failed to respond to standard systemic therapy, or for whom standard or curative systemic therapy does not exist, is not tolerable or was refused
* Patients should be at least 4 weeks from last receipt of a cytotoxic or biological agent prior to start of SBRT, with the exception of mitomycin C which requires a 6-week washout
* Patients should have unresectable disease or not be a candidate for surgical resection
* Patients must have a minimum of 1 and a maximum of 5 separate metastatic lesions planned for SBRT. (Patients may have > 5 metastatic lesions overall, however only up to 5 lesions will be treated with SBRT.) SBRT sites must be equal to or less than 5 cm in greatest dimension. SBRT treated sites must be measurable per RECIST 1.1 and can include metastatic sites in the lung, liver, or soft tissue. Sites that are intracranial or in the bone are excluded. Sites deemed not appropriate for SBRT by the treating radiation oncologist are also excluded
* Patients should be at least 4 weeks from last radiation therapy prior to starting SBRT
* Patients should be at least 4 weeks from any investigational therapy prior to starting SBRT, with the exception of prior immunotherapy which would require a 3 month washout
* Patients should have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patients should be considered clinically stable with an estimated overall survival of at least 3 months
* Neutrophil count > 1500/mm^3
* Lymphocyte count > 500/mm^3
* Hemoglobin > 9 gm/dl
* Platelets count > 100,000/mm^3
* Aspartate transaminase (AST)/alanine transaminase (ALT) < 2.5 x upper limit of normal (ULN)
* Bilirubin ≤ ULN
* Patients should have adequate kidney function defined as a serum creatinine < ULN or calculated creatinine clearance of > 60ml/min (Cockroft-Gault formula)
* Patients should have adequate cardiac function defined as:

  * No history of acute coronary syndromes (including myocardial infarction, unstable angina, Coronary artery bypass grafting (CABG), coronary angioplasty, or stenting) < 12 months prior to screening
  * No impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:

    * Symptomatic chronic heart failure;
    * Evidence of clinically significant cardiac arrhythmias and/or conduction abnormalities
  * No uncontrolled arterial hypertension despite appropriate medical therapy (defined as systolic blood pressure > 160 or diastolic blood pressure >100)
  * Electrocardiogram (EKG) showing normal sinus rhythm and a corrected QT (QTc) ≤ 450 ms for male and ≤ 470 ms for female patients
* Patients should have adequate pulmonary function defined as:

  * Lack of uncontrolled pleural effusion requiring recurrent draining procedures (more than once per month)
  * Lack of oxygen supplementation dependence
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Screening 2-dimensional (2-D) echocardiogram (echo) shows a left ventricular ejection fraction (LVEF) > 40%
* Urinalysis shows lack of proteinuria or a maximum of 1+ proteinuria
* Women of childbearing potential should use highly effective contraception while receiving the trial regimen and for at least 5 half-lives of M5A-IL2 from the last dose of M5A-IL2

Exclusion Criteria:

* Patients on immunosuppressive treatments including supra-physiological doses of corticosteroids
* Patients with history of auto-immune disease including history of inflammatory bowel disease
* Patients with active brain metastases
* Patients in the child-bearing ages who refuse to use adequate birth control measures (example: contraceptives, barrier method, or abstinence)
* Lactating females who do not agree to stop breastfeeding
* Known active hepatitis B or C
* Major surgical procedure within 4 weeks prior to SBRT
* Non-healed wound or surgical incisions
* Radiographic evidence of bowel obstruction
* Electrolyte disturbances (sodium, potassium, magnesium, calcium, and phosphorous) that are not correctable to at least CTCAE grade 1 with replacement therapy
* Known hypersensitivity of any of the study drug agents or components
* Patients should not have any uncontrolled illness including ongoing or active infection
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study agents
* Pregnant women are excluded from this study because the investigational agents on this study are highly likely to exert teratogenic or abortifacient effects
* Patients with other active malignancies are ineligible for this study
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-09-05 (Estimated); Study Completion 2026-09-05 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of the M5A-IL2 immunocytokine (M5A-ICK) | At the end of cycle 1 (each cycle is 28 days)
  Will be assessed following accelerated titration design 3, single patient cohorts will be used with dose doubling between cohorts until either a dose limiting toxicity (DLT) is observed, or 2 patients experience a moderate (grade 2) M5A-ICK related adverse event. At dose level 5, the design reverts to 3 patient cohorts (following the traditional 3+3 design) with 40% increments between dose levels. In the traditional 3+3 design, once 3 patients at a dose level are evaluable, if none has experienced a DLT, the dose can be escalated.
Recommended phase 2 dose | At the end of cycle 1 (each cycle is 28 days)
  Will either be the MTD, or below, based on the full consideration of late adverse events, sub-DLT toxicities, clinical activity, and biological correlatives.

SECONDARY OUTCOMES:
Therapeutic response to treatment | Up to 2 years
  Will be reported according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Incidence of adverse events | Up to 3 months after last M5A-ICK injection
  All adverse events, including allergic reactions, hypertension, hypotension, and infusion reactions will be summarized in terms of dose level, type and frequency, data of onset and duration (where relevant) using Common Terminology Criteria for Adverse Events [CTCAE] version 5.0.
Number of participants with treatment-related auto-antibody formation | Screening, days 8 and 36, and 3 months
  Frequency of participants with auto-antibody formation, overall and by dose of M5A-IL2.
Pharmacokinetics of M5A-IL2 (M5A-ICK blood clearance ) | Pre-injection, approximately 1, 4 and 6 hours post injection on each day, and one sample done 1 and 2 days following the 3rd subcutaneous dose of M5A-IL2
  Blood samples up to 4 days (based on the predicted ICK half life of 10 hours) will be used to determine M5A-ICK blood clearance by ELISA analysis using human CEA for capture and reporting with anti-IL2-HRP.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Y Wong, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States